CLINICAL TRIAL: NCT00481338
Title: Knee and Hip OsteoArthritis Long Term Assessment. Prevalence, Natural History, Prognosis Factor, Quality of Life, Health Care Consumption and Social Consequences of Symptomatic Knee and Hip Osteoarthritis in France
Brief Title: Prevalence,Natural History,Prognosis Factor,QualityofLife,Health Care Consumption and Social Consequences of Symptomatic Knee and Hip Osteoarthritis in France
Acronym: KHOALA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DGS2006-0146
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: Cohort; Quality of life; Health resource use; Disability; Prognosis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study specific procedure (Experimental): X-rays, biological samples and medical information about osteoarthritis
  Interventions: Procedure: X-rays; Biological: biological samples; Other: medical information about osteoarthritis

INTERVENTIONS:
Procedure: X-rays — X-rays (hip and knee) every 2 years
Biological: biological samples — biological sample (blood and urine) every 2 years
Other: medical information about osteoarthritis — several questionnaires about pain and function (WOMAC), physical activity (MAQ), quality of life (generic SF-36 and OA specific OAKHQOL/AMIQUAL), comorbidities (FCI), mental status (MMS), heath status (GHQ 28) and health resource consumption

SUMMARY:
The aim of the project is to assemble and to follow on a 10-year period a nationwide representative sample of lower limb OA patients.

General objectives: To document the natural history and to identify predictive factors of the evolution and consequences of hip and knee OA in terms of pain, functional disability, structural damage, quality of life, autonomy, medical and health care use and cost of disease.

ELIGIBILITY:
Inclusion Criteria:

* male and female aged between 40 and 75 years
* symptomatic hip or knee, uni or bilateral OA with clinical diagnosis confirmed by a medical physician and satisfying ACR classification criteria
* Representative of prevalent cases in France at the cohort set-up time

Exclusion Criteria:

* presence of hip or knee joint replacement surgery
* comorbidities severe enough to affect quality of life significantly or likely to induce a high health care consumption independently of OA
* an history of osteotomy
* Patello-femoral osteoarthritis without tibio-femoral osteoarthritis
* Other joint diseases of the target joints
* adult under legal protection or not able to consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2007-04; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Quality of life, patient reported outcome measures | every year, up to 10 years

SECONDARY OUTCOMES:
health care consumption | every year, up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Francis Guillemin, MD, PhD, Principal Investigator — CHU Nancy (promoteur)
Locations (6):
- France (6):
  - Patrice Fardellone, Amiens
  - CHU de la Cavale Blanche, Brest
  - CHU Nancy, hopital brabois, Nancy
  - CHU l'Archet, Nice
  - Hôpital de la Pitié-Salpêtrière, Paris
  - CHU Rangueil, Toulouse

REFERENCES:
- [Derived] Garnero P, Guillemin F, Ngueyon Sime W, Gineyts E, Chapurlat R, Roux C. Cartilage turnover, but not novel synovial collagen marker, is associated with joint damage progression in osteoarthritis patients. Rheumatology (Oxford). 2025 Sep 26:keaf510. doi: 10.1093/rheumatology/keaf510. Online ahead of print. PMID 41002273